CLINICAL TRIAL: NCT03986307
Title: The Effect of Omega-3 Supplementation on Muscle Functioning, Inflammation and Muscle Signaling in Elderly
Brief Title: The Effect of Omega-3 Supplementation on Muscle Functioning, Inflammation and Muscle Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, sebastiaan dalle, Doctoral researcher, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S61809
Record Dates: First submitted 2019-06-04; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Aging
Keywords: muscle metabolism; inflammation; muscle molecular signaling; muscle functioning
MeSH Terms: conditions — Inflammation | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Elderly humans (>65y) are randomized to a placebo or omega-3 group (interventions, tests, analyses etc. are executed in parallel).
Who Masked: Participant, Investigator
Masking Description: Subjects are a priori randomized to one of both conditions. Both groups undergo an identical intervention, but receive different supplements (although appearance-matched). The investigators do not know in which condition the subjects are randomized. One researcher, who is not involved in the intervention/data collection/data analyses, holds the code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Experimental): Elderly supplemented with omega-3.
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acid supplementation; Other: Resistance exercise
- Placebo (Placebo Comparator): Elderly supplemented with corn oil.
  Interventions: Other: Resistance exercise; Dietary Supplement: Placebo - appearance-matched oil supplementation

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acid supplementation — Daily supplementation with omega-3 capsules (daily for 14 weeks). Each day: 3 capsules of 1.1g
  Arms: Omega-3
Other: Resistance exercise — Resistance exercise training in both supplementation conditions (3 times per week for 12 weeks).
Dietary Supplement: Placebo - appearance-matched oil supplementation — Daily supplementation with placebo capsules (daily for 14 weeks). Each day: 3 capsules of 1.1g
  Arms: Placebo

SUMMARY:
Elderly are supplemented with either Omega-3 (3 x 1.1g per day) or placebo (corn oil) during 14 weeks. The last 12 weeks, supplementation is combined with resistance exercise training (3x per week) focusing on upper leg strength. In the present project, the investigators study whether differences in muscle strength and/or muscle mass between conditions can be explained by omega-3-induced effects on systemic or muscle inflammatory signaling, or differences in muscle molecular signaling.

DETAILED DESCRIPTION:
Elderly are supplemented with either Omega-3 (3 x 1.1g per day) or placebo (corn oil) during 14 weeks. The last 12 weeks, supplementation is combined with resistance exercise training (3x per week) focusing on upper leg strength. In the present project, the investigators study whether differences in muscle strength and/or muscle mass between conditions can be explained by omega-3-induced effects on systemic or muscle inflammatory signaling, or differences in muscle molecular signaling.

ELIGIBILITY:
Inclusion Criteria:

* aged >= 65 years

Exclusion Criteria:

* BMI < 20; BMI > 35
* regular NSAID intake in the last 3 months
* omega-3 supplementation in the last year
* regular resistance exercise in the last year
* cancer, liver and renal disease, unstable cardiovascular disease, musculoskeletal disease
* cognitive limitations that might interfere with the (adherence to) the intervention or with the testing of outcome parameters
* unstable body weight
* smoking

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Isometric muscle strength | Change in muscle strength between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Isometric muscle strength as assessed with Biodex Device in Nm
Systemic inflammatory signaling | Change in inflammatory signaling between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Systemic (blood) markers of inflammation: hs-CRP (mg/L), IL-6 (pg/mL), TNFa (pg/mL)
Muscle strength | Change in muscle strength between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  One Repetition Maximum on the leg press fitness device in kg

SECONDARY OUTCOMES:
Muscle quality | Change in muscle quality between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  muscle strength (Torque) per muscle volume
Muscle molecular signaling (Protein levels of anabolic/catabolic signaling and skeletal muscle stress) | Change in muscle molecular signaling between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Biochemical analyses of muscle biopsies obtained pre-post intervention in both conditions.
  This involves parameters of muscle anabolism, catabolism, stress, structure, integrity, quality etc.: mTORC1 pathway, FoXO, MAPK (western blotting technique, values expressed as arbitrary units)

OTHER OUTCOMES:
Handgrip strength | Change in handgrip strength between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Handgrip strength measured by a dynamometer (results in kg)
Timed up-and-go test | Change in timed up-and-go test performance between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Timed-up-and-go: time needed to stand up from a chair, walk 3m, turn, walk back and sit down.
Sit-to-stand test | Change in sit-to-stand test performance between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Sit-to-stand: the amount of repetitions that one can complete during 30 sec and the time needed to complete 5 sit-to-stands.
Fat% | Change in fat% between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Bioelectrical impedance analysis-derived fat %
Lean mass% | Change in lean mass% between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Bioelectrical impedance analysis-derived lean mass %
Basal metabolic rate | Change in basal metabolic rate between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Bioelectrical impedance analysis-basal metabolic rate (kcal)
Muscle Volume Left | Change in muscle volume between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Muscle Volume in a 2-cm CT-scan slice (4 slices of 5mm)
Mean Muscle Hounsfield Unit | Change in Mean Muscle Hounsfield Unit between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Muscle Hounsfield Unit serves as a marker of muscle quality
Sleep | Change in sleep quality between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Questionnaire (Pittsburgh Sleep Quality Index)
Stress | Change inperceived stress between prior to and following the study intervention of 14 weeks (Jan - May 2019)
  Questionnaire (Perceived Stress Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No